CLINICAL TRIAL: NCT01297062
Title: A Randomized, Phase 1, Three-Period, Placebo- and Positive-Controlled, Double-Blind, Crossover Study to Assess the Electrophysiological Effects of Exenatide at Therapeutic and Supratherapeutic Concentrations on the 12-Lead Electrocardiogram QT Interval in Healthy Subjects
Brief Title: A Safety Study to Assess the Effects of Therapeutic and Supratherapeutic Exenatide Concentrations on QT Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: BCB112
Record Dates: First submitted 2011-02-09; First posted 2011-02-16 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Subjects
Keywords: Diabetes; exenatide; Amylin; Lilly; QT interval
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exenatide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo comparator
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Exenatide — IV Exenatide (therapeutic and supratherapeutic concentrations)
  Arms: Exenatide
Drug: Moxifloxacin — Oral Moxifloxacin (400 mg)
  Arms: Moxifloxacin
Drug: Placebo comparator — IV Placebo (matching volume of placebo)
  Arms: Placebo

SUMMARY:
Compare the effect of exenatide (therapeutic and supratherapeutic concentrations), moxifloxacin and placebo on the QT interval.

ELIGIBILITY:
Inclusion Criteria:

* Is overtly healthy, as determined by medical history and physical examination
* Has body mass index (BMI) between 25 and 35 kg/m2
* Has fasting serum glucose <110 mg/dL
* Has no clinically significant blood pressure or heart rate readings as judged by the investigator at study start
* Has electrocardiogram (ECG) results judged as not clinically significant by the investigator at study start

Exclusion Criteria:

* Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being
* Has an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as a Bazett's corrected QT (QTcB) interval >450 ms.
* Family history of sudden death
* Personal history of unexplained syncope within last year, or family history of Long QT Syndrome, or significant active cardiac disease, or symptoms of angina pectoris or transient ischemic attacks within the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Research and Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (2):
- United States (2):
  - Research Site, Daytona Beach, Florida
  - Research Site, Evansville, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Exenatide-Moxifloxacin Sequence: Placebo comparator in Period I; Exenatide in Period II; Moxifloxacin with placebo infusion in Period III;
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Exenatide-Moxifloxacin-Placebo Sequence: Exenatide in Period I; Moxifloxacin with placebo infusion in Period II; Placebo comparator in Period III
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Moxifloxacin-Placebo-Exenatide Sequence: Moxifloxacin with placebo infusion in Period I; Placebo comparator in Period II; Exenatide in Period III
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Moxifloxacin-Exenatide-Placebo Sequence: Moxifloxacin with placebo infusion in Period I; Exenatide in Period II; Placebo comparator in Period III
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Placebo-Moxifloxacin-Exenatiden Sequence: Placebo comparator in Period I; Moxifloxacin with placebo infusion in Period II; Exenatide in Period III
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Exenatide-Placebo-Moxifloxacin Sequence: Exenatide in Period I; Placebo comparator in Period II; Moxifloxacin with placebo infusion in Period III
  Exenatide - stepped intravenous (IV) infusion to gradually deliver levels of exenatide at concentrations of approximately 200 pg/mL (Day 1), 300 pg/mL (Day 2), and 500 pg/mL (Day 3)
  Moxifloxacin - Placebo intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) with single oral dose of Moxifloxacin (400 mg) on Day 2
  Placebo - intravenously infused at the same volume rate (mL/min) as that of active study medication (exenatide) on Day 1, Day 2, and Day 3
- Non-Randomized: Not Randomized
Period: Overall Study
Arm/Group | Placebo-Exenatide-Moxifloxacin Sequence | Exenatide-Moxifloxacin-Placebo Sequence | Moxifloxacin-Placebo-Exenatide Sequence | Moxifloxacin-Exenatide-Placebo Sequence | Placebo-Moxifloxacin-Exenatiden Sequence | Exenatide-Placebo-Moxifloxacin Sequence | Non-Randomized
Started | 15 | 14 | 14 | 14 | 15 | 14 | 8
Intent to Treat (ITT) | 15 | 14 | 14 | 14 | 15 | 14 | 0
Evaluable Population | 11 | 12 | 12 | 13 | 13 | 13 | 0
Completed | 11 | 13 | 12 | 13 | 13 | 13 | 0
Not Completed | 4 | 1 | 2 | 1 | 2 | 1 | 8
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Decision | 1 | 1 | 0 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo-Exenatide-Moxifloxacin Sequence: Placebo comparator in Period I; Exenatide in Period II; Moxifloxacin with placebo infusion in Period III
- Exenatide-Moxifloxacin-Placebo Sequence: Exenatide in Period I; Moxifloxacin with placebo infusion in Period II; Placebo comparator in Period III
- Moxifloxacin-Placebo-Exenatide Sequence: Moxifloxacin with placebo infusion in Period I; Placebo comparator in Period II; Exenatide in Period III
- Moxifloxacin-Exenatide-Placebo Sequence: Moxifloxacin with placebo infusion in Period I; Exenatide in Period II; Placebo comparator in Period III
- Placebo-Moxifloxacin-Exenatiden Sequence: Placebo comparator in Period I; Moxifloxacin with placebo infusion in Period II; Exenatide in Period III
- Exenatide-Placebo-Moxifloxacin Sequence: Exenatide in Period I; Placebo comparator in Period II; Moxifloxacin with placebo infusion in Period III
- Total: Total of all reporting groups
Arm/Group | Placebo-Exenatide-Moxifloxacin Sequence | Exenatide-Moxifloxacin-Placebo Sequence | Moxifloxacin-Placebo-Exenatide Sequence | Moxifloxacin-Exenatide-Placebo Sequence | Placebo-Moxifloxacin-Exenatiden Sequence | Exenatide-Placebo-Moxifloxacin Sequence | Total
Number analyzed (Participants) | 15 | 14 | 14 | 14 | 15 | 14 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (8.98) | 45.1 (11.43) | 43.7 (11.56) | 37.8 (10.66) | 43.3 (13.74) | 41.0 (10.50) | 42.1 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 0 | 2 | 1 | 8
  Male | 15 | 12 | 11 | 14 | 13 | 13 | 78
Weight [Mean (Standard Deviation); unit: kilogram] | 87.66 (8.107) | 81.16 (11.235) | 90.77 (12.375) | 93.66 (11.704) | 89.71 (7.726) | 90.71 (11.251) | 88.94 (10.899)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Least Squares (LS) Mean Changes From Baseline in Population-based Corrected QT Intervals (QTcP) Between Exenatide and Placebo on Day 1 Averaged Over 1300h, 1400h, 1500h (Target Steady State Exenatide Concentration of 200 pg/mL)
Description: Factors in QT correction formulas were first estimated using pre-therapy data. The most appropriate correction method (QTcP) minimized the mean squared individual QTc/RR regression slope with on-exenatide data. Adequacy of correction was validated with on-placebo data. Change from baseline in QTcP was analyzed by a mixed-effects model for repeated measures (MMRM) between exenatide and placebo.
Time Frame: Baseline, Day 1
Population: Evaluable Population included all ITT subjects who completed all ECG assessment periods and have valid ECG measurements and no vomiting in any ECG data extraction window. No missing value was imputed.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Exenatide: Exenatide
- Placebo: Placebo Comparator
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 74 | 74
msec | -2.25 (0.636) [-3.30 to -1.20] | -0.89 (0.599) [-1.88 to 0.10]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; 60 evaluable subjects gives more than 90% power to show non-inferiority of exenatide versus placebo, using t-test in 2-way crossover, alpha=0.05, true difference of 5 msec, and standard deviation of the within-subject difference of 10.04 msec; Test type: Non-Inferiority or Equivalence — Non-inferiority is established if the upper limit of 2-sided 90% confidence interval (CI), equivalent to the upper limit of 1-sided 95% CI, for change from baseline in QTcP (exenatide - placebo) is below 10 msec; Mixed Models Analysis — No adjustment on CI for the primary outcome measure; Least Squares Mean Difference = -1.36, 90% CI 2-sided [-2.21 to -0.50] — The MMRM includes Treatment (Exenatide versus Placebo), Day, Time, Period, Sequence, and Day-Time-Treatment interaction as fixed effects, subject random intercept

2. Primary Outcome: Comparison of LS Mean Changes From Baseline in QTcP Intervals Between Exenatide and Placebo on Day 2 Averaged Over 1300h, 1400h, 1500h (Target Steady State Exenatide Concentration of 300 pg/mL)
Description: Factors in QT correction formulas were first estimated using pre-therapy data. The most appropriate correction method (QTcP) minimized the mean squared individual QTc/RR regression slope with on-exenatide data. Adequacy of correction was validated with on-placebo data. Change from baseline in QTcP was analyzed by a MMRM between exenatide and placebo.
Time Frame: Baseline, Day 2
Population: Evaluable Population. No imputation for missing value was used.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 74 | 74
msec | -2.58 (0.640) [-3.64 to -1.52] | -0.56 (0.596) [-1.54 to 0.43]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority is established if the upper limit of 2-sided 90% CI, equivalent to the upper limit of 1-sided 95% CI, for change from baseline in QTcP (exenatide - placebo) is below 10 msec; Mixed Models Analysis — No adjustment on CI for the primary outcome measure; Least Squares Mean Difference = -2.02, 90% CI 2-sided [-2.88 to -1.16] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Comparison of LS Mean Changes From Baseline in QTcP Intervals Between Exenatide and Placebo on Day 3 Averaged Over 1300h, 1400h, 1500h (Target Steady State Exenatide Concentration of 500 pg/mL)
Description: as for outcome 2
Time Frame: Baseline, Day 3
Population: Evaluable Population. No imputation for missing value was used.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 74 | 74
msec | -3.54 (0.675) [-4.66 to -2.42] | -2.41 (0.623) [-3.44 to -1.38]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis — No adjustment on CI for the primary outcome measure; Least Squares Mean Difference = -1.13, 90% CI 2-sided [-2.11 to -0.15] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Assay Sensitivity of Moxifloxacin at 1000h (1 Hour Post-administration of Moxifloxacin) on Day 2
Description: Change from baseline in QTcP was analyzed by a MMRM between moxifloxacin and placebo.
Time Frame: Baseline, Day 2
Population: Evaluable Population. No imputation for missing value was used.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Moxifloxacin: Moxifloxacin with placebo infusion
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 74 | 74
msec | 1.91 (1.079) [0.12 to 3.70] | -3.56 (0.953) [-5.14 to -1.98]
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; Assay sensitivity of moxifloxacin is established if the lower limit of the 2-sided 90% CI for difference in change from baseline in QTcP (moxifloxacin - placebo) is greater than 5 msec; Test type: Superiority or Other; Mixed Models Analysis; Least Squares Mean Difference = 5.47, 90% CI 2-sided [2.82 to 8.12] — The MMRM includes Treatment (Moxifloxacin versus Placebo), Time, Period, Sequence, and Time-Treatment interaction as fixed effects, subject random intercept. Multiplicity adjusted CI for the mean difference is shown

5. Secondary Outcome: Assay Sensitivity of Moxifloxacin at 1100h (2 Hour Post-administration of Moxifloxacin) on Day 2
Description: Change from baseline in QTcP was analyzed by a MMRM between moxifloxacin and placebo.
Time Frame: Baseline, Day 2
Population: Evaluable Population. No imputation for missing value was used.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 74 | 74
msec | 9.75 (0.934) [8.20 to 11.30] | -0.81 (0.872) [-2.26 to 0.63]
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Least Squares Mean Difference = 10.56, 90% CI 2-sided [8.46 to 12.67] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Assay Sensitivity of Moxifloxacin at 1200h (3 Hour Post-administration of Moxifloxacin) on Day 2
Description: Change from baseline in QTcP was analyzed by a MMRM between moxifloxacin and placebo.
Time Frame: Baseline, Day 2
Population: Evaluable Population. No imputation for missing value was used.
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 74 | 74
msec | 12.47 (1.011) [10.79 to 14.15] | 1.56 (0.828) [0.18 to 2.93]
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Least Squares Mean Difference = 10.92, 90% CI 2-sided [8.71 to 13.13] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Number of Subjects With QTcP Interval >450msec at Any Timepoint on Any Day in Exenatide and Placebo
Description: Number of subjects with QTcP > 450 msec at any timepoint on any day was summarized by frequency for exenatide and placebo.
Time Frame: Day 1, 2, or 3
Population: Evaluable Population. No imputation for missing value was used.
Measure: Number; unit: participants
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 74 | 74
participants | 0 | 0

8. Secondary Outcome: Number of Subjects With Increase of QTcP Interval From Baseline >30msec at Any Timepoint on Any Day in Exenatide and Placebo
Description: Number of subjects with increase of QTcP interval from baseline >30 msec at any timepoint on any day was summarized by frequency for exenatide and placebo.
Time Frame: Baseline, Day 1, 2, or 3
Population: Evaluable Population. No imputation for missing value was used.
Measure: Number; unit: particpants
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 74 | 74
particpants | 0 | 0

9. Secondary Outcome: Plasma Exenatide Concentrations at Steady State on Day 1, 2 and 3
Description: The plasma exenatide concentration at steady state was descriptively summarized by geometric mean, standard error, and its effect on placebo-adjusted change from baseline in QTcP was assessed.
Time Frame: Baseline, Day 1, 2, and 3
Population: Evaluable Population. No imputation for missing value was used. Day 1, 2, and 3 exenatide concentration < LLOQ was set to missing.
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Exenatide
Number analyzed (Participants) | 68
pg/mL
  Day 1 | 252.74 (8.454)
  Day 2 | 399.14 (11.936)
  Day 3 | 626.65 (21.159)
Statistical Analysis 1: Comparison: Exenatide; The analysis is to test the significance of the linear regression slope (null hypothesis: slope equal to zero) between placebo-adjusted change from baseline in QTcP and exenatide concentration; Test type: Superiority or Other; p = 0.5962, Mixed Models Analysis; Slope = 0.0008, 90% CI 2-sided [-0.0017 to 0.0033] — The linear mixed-effects model includes placebo-adjusted change from baseline in QTcP as response, plasma exenatide concentration as covariate, fixed intercept of zero, subject random slope

ADVERSE EVENTS:
Arm/Group | Exenatide | Placebo | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/84 | 1/80
Other Adverse Events (participants affected / at risk) | 65/80 | 10/84 | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=80) | Placebo (N=84) | Moxifloxacin (N=80)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=80) | Placebo (N=84) | Moxifloxacin (N=80)
NAUSEA (Gastrointestinal disorders) | 36 | 1 | 2
VOMITING (Gastrointestinal disorders) | 23 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 18 | 3 | 2
HEADACHE (Nervous system disorders) | 16 | 6 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 15 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 14 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 8 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 7 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 7 | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 0 | 0
DIZZINESS (Nervous system disorders) | 6 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 4 | 0 | 1
EARLY SATIETY (General disorders) | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less